CLINICAL TRIAL: NCT01199042
Title: BiPAP (Automatic Servo Ventilation) autoSV Advanced in Central Apnea Patients
Brief Title: Bipap Automatic Servo Ventilation (autoSV) Advanced in Central Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-1001-ASVWO-MS
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Cheyne-Stokes Respiration; Sleep Apnea, Central
MeSH Terms: conditions — Cheyne-Stokes Respiration; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BiPAP autoSV Advanced Device (Other): Positive airway pressure device
  Interventions: Device: BiPAP autoSV Advanced

INTERVENTIONS:
Device: BiPAP autoSV Advanced — The sleep apnea device will be set-up in automatic mode with the settings wide open for the entire night.

SUMMARY:
Pilot study testing the Bipap autoSV Advanced Algorithm during full night, in-lab polysomnography (PSG) and 3 months at home on patients with Central Sleep Apnea, Hunter Cheyne Stokes Respiration, or Complex Sleep Apnea.

DETAILED DESCRIPTION:
Participants who qualify will be scheduled for one full night, attended diagnostic PSG, one full night attended continuous positive airway pressure (CPAP) titration, and one full night attended BiPAP autoSV Advanced titration PSG. Participants will be provided a BiPAP autoSV Advanced to use at home for 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 21-75.
2. Able and willing to provide written informed consent.
3. Diagnosis of Central Sleep Apnea such as Hunter Cheyne Stokes Breathing, Complex Sleep Apnea, or Central Apnea with current daily Opioid use or any other predominant central sleep apnea.

   1. For participants diagnosed with Hunter Cheyne Stokes Breathing, at least 3 cycles of crescendo-decrescendo breathing amplitude AND either a Central Apnea Index (CAI) ≥ 5/hour OR the crescendo-decrescendo cycles last at least 10 consecutive minutes from an attended Diagnostic Polysomnogram (PSG).
   2. For participants diagnosed with Central Sleep Apnea with current daily Opioid use or any other predominant central sleep apnea, an Apnea/Hypopnea Index (AHI) ≥ 15 and CAI > 5 from an attended Diagnostic PSG.
   3. For participants diagnosed with Complex Sleep Apnea, an AHI ≥ 15 and CAI > 5 from a CPAP titration.
4. Systolic blood pressure > 80 mm Hg at Visit 1.
5. Agreement to undergo a full-night, attended Diagnostic PSG.
6. Agreement to undergo a full-night, attended CPAP titration PSG.
7. Agreement to undergo a full-night, attended BiPAP automatic Servo Ventilation (autoSV) Advanced titration PSG

Exclusion Criteria:

1. Active participation in another interventional research study.
2. Diagnosis of acute decompensated heart failure.
3. Surgery of the upper airway, nose, sinus or middle ear within the last 90 days.
4. Major medical or psychiatric condition that would interfere with the demands of the study or the ability to complete the study. For example, severe unstable chronic lung disease, neuromuscular disease, cancer, or end stage renal failure.
5. Qualifying for or awaiting heart transplantation.
6. Currently prescribed oxygen therapy (e.g. as needed, nocturnal, or continuous).
7. At home treatment with adapted Servo Ventilation (ASV) or Bilevel Positive Airway Pressure (PAP) therapies.
8. Unable to use PAP therapies due to physical (e.g. facial structural abnormalities) or cognitive (e.g. dementia) issues.
9. Participants in whom PAP therapy is medically contraindicated.
10. Uncontrolled hypertension (systolic ≥ 200 mm Hg/diastolic ≥ 120 mm Hg).
11. Narcolepsy.
12. Untreated Restless Legs Syndrome.
13. Periodic Limb Movement arousal index > 20/hr.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh Javaheri, MD, Principal Investigator — Sleepcare Diagnostics
Locations (3):
- United States (3):
  - Gaylord Hospital - Gaylord Sleep Research, Wallingford, Connecticut
  - Kentucky Research Group, Louisville, Kentucky
  - Sleepcare Diagnostics, Mason, Ohio

REFERENCES:
- [Derived] Javaheri S, Winslow D, McCullough P, Wylie P, Kryger MH. The Use of a Fully Automated Automatic Adaptive Servoventilation Algorithm in the Acute and Long-term Treatment of Central Sleep Apnea. Chest. 2015 Dec;148(6):1454-1461. doi: 10.1378/chest.14-2966. PMID 25950507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-nine patients were enrolled between September 2010 and February 2013. Two participants did not meet) criteria after centralized scoring of diagnostic and CPAP polysomnograms (PSGs) and were excluded from analysis. Twenty-seven participants (five women) completed 3 nights in-laboratory attended PSG, and 26 completed 3 months of follow-up.
Groups:
- Diagnostic, Continuous Positive Airway Pressure (CPAP), ASV: All participants first underwent a full night, attended diagnostic PSG. Eligible participants then had an attended full night Continuous Positive Airway Pressure (CPAP) manual titration followed by full night, attended, but automated titration with the BiPAP automatic Servo Ventilation.(AutoSV) Advanced™ (Philips Respironics, Murrysville, PA), device.
Period: Sleep Laboratory (3 Nights)
Arm/Group | Diagnostic, Continuous Positive Airway Pressure (CPAP), ASV
Started | 29
Completed | 27
Not Completed | 2
Not completed — Didn't meet inclusion/exclusion criteria | 2
Period: At Home (3 Months)
Arm/Group | Diagnostic, Continuous Positive Airway Pressure (CPAP), ASV
Started | 27
Completed | 26
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Diagnostic, Then CPAP, Then BiPAP autoSV Advanced: Diagnostic, then CPAP, then BiPAP autoSV Advanced (within-subjects design)
Arm/Group | Diagnostic, Then CPAP, Then BiPAP autoSV Advanced
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 1
  Caucasian | 25
  African American, Irish, Native American | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Apnea/Hypopnea Index (AHI)
Description: To compare the AHI between the diagnostic CPAP titration and BiPAP autoSV Advanced PSG nights.
Time Frame: During a single night of polysomnography lasting up to 8 hours.
Measure: Mean (Standard Deviation); unit: Apnea-Hypopnea events per hour
Groups:
- Diagnostic Apnea-Hypopnea Index: Participants had Diagnostic PSG where the Apnea-Hypopnea Index was measured
- Continuous Positive Airway Pressure Apnea-Hypopnea Index: The CPAP machine was used to determine the Apnea-Hypopnea Index.
- BiPAP autoSV Apnea-Hypopnea Index: The BiPAP autoSV machine was used to determine the Apnea-Hypopnea Index
Arm/Group | Diagnostic Apnea-Hypopnea Index | Continuous Positive Airway Pressure Apnea-Hypopnea Index | BiPAP autoSV Apnea-Hypopnea Index
Number analyzed (Participants) | 27 | 27 | 27
Apnea-Hypopnea events per hour | 55 (24) | 37 (22) | 12 (20)

2. Secondary Outcome: Epworth Sleepiness Scale
Description: To determine if there are changes in subjective sleepiness on the Epworth Sleepiness Scale (ESS) between Baseline (Visit 1) and 3 months (Visit 6). The ESS is an 8 question survey that determines sleepiness, each question is rated as a 0-3 will the total score ranging from 0-24.
  Interpretation:
  Score 0-7: Unlikely that there is abnormal sleep Score 8-9: Average amount of daytime sleepiness Score 10-15: Possible excessive sleepiness depending on the situation. Patient may want to consider seeking medical attention.
  Score 16-24: Excessive sleepiness and patient should consider seeking medical attention
  A decrease in the score indicates improvements in a patients overall sleepiness. An increase in the score indicates increased sleepiness.
Time Frame: 3 months
Population: 26 participants completed the 3-month home follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BiPAP autoSV Advanced Device: Over the 90-day home treatment period, the Auto-Servo Ventilation (ASV) device consistently treated obstructive and central Sleep Disordered Breathing (SDB) events.
Arm/Group | BiPAP autoSV Advanced Device
Number analyzed (Participants) | 26
units on a scale
  Baseline (visit 1) | 12.8 (5)
  3 months (visit 6) | 7.8 (4)

3. Secondary Outcome: Breathing Event Indexes
Description: To determine if there are changes in breathing event indexes (Encore Pro Software) from the first 7 days of BiPAP autoSV Advanced at home treatment to the last 7 days of at home treatment to assess therapy efficacy.
  Values were determined by taking the average of the first 7 days of treatment and comparing them to the average of the last 7 days of treatment.
Time Frame: from the first 7 days of BiPAP autoSV Advanced at home treatment to the last 7 days of at home treatment
Population: 26 participants completed the 3-month home follow-up.
Measure: Mean (Standard Deviation); unit: Apnea-Hypopnea events per hour
Arm/Group | BiPAP autoSV Advanced Device
Number analyzed (Participants) | 26
Apnea-Hypopnea events per hour
  First Week | 11.6 (8.7)
  Last Week | 10.0 (6.8)

4. Secondary Outcome: Average Therapy Pressure Values
Description: To compare BiPAP autoSV Advanced therapy pressure values (Encore Pro Software) from the first 7 days of BiPAP autoSV Advanced at home treatment to the last 7 days of at home treatment to determine if pressure requirements change over time.
  This analysis compares the average pressure support of the first week compared to the average pressure support to the final week.
Time Frame: 3 months
Population: 26 participants completed the 3-month home follow-up.
Measure: Mean (Standard Deviation); unit: cm/H2O
Arm/Group | Diagnostic, Continuous Positive Airway Pressure (CPAP), ASV
Number analyzed (Participants) | 26
cm/H2O
  First Week | 3.7 (2.0)
  Last Week | 3.9 (1.7)

ADVERSE EVENTS:
Time Frame: Duration of study: 2 years and 5 months
Groups:
- Diagnostic, Then CPAP, Then BiPAP autoSV Advanced: Participants had a diagnostic PSG, then CPAP and BiPAP autoSV. Participants then went home and used the autoSV for 90 days.
Arm/Group | Diagnostic, Then CPAP, Then BiPAP autoSV Advanced
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No